CLINICAL TRIAL: NCT06866691
Title: Comparison of Levetiracetam Versus Lacosamide for Seizure Prevention in Moderate to Severe Traumatic Brain Injured Patients
Brief Title: Seizure Prevention in Traumatic Brain Injury With Levetiracetam and Lacosamide
Acronym: SEIZE-TBI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00123210
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injury; Post-Traumatic Seizures; Seizure Medication
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Levetiracetam; Lacosamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- levetiracetam (Experimental): levetiracetam 1000 mg intravenously or by mouth twice daily for a total of 7 days
  Interventions: Drug: levetiracetam
- lacosamide (Experimental): lacosamide 200 mg intravenously or by mouth twice daily for a total of 7 days
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: levetiracetam — levetiracetam 1000 mg intravenously or by mouth twice daily for a total of 7 days
  Other Names: Keppra
  Arms: levetiracetam
Drug: lacosamide — lacosamide 200 mg intravenously or by mouth twice daily for a total of 7 days
  Other Names: Vimpat
  Arms: lacosamide

SUMMARY:
The purpose of this study is to assess the incidence of early post-traumatic seizures. The study will also assess the benefit of lacosamide compared to levetiracetam in regards to agitation and behavioral adverse effects in patients with moderate to severe traumatic brain injury requiring seizure prophylaxis.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial of patients with moderate to severe TBI requiring seizure prophylaxis to prevent early and late posttraumatic seizures. Patients will be identified and randomized as soon as possible, within 24 hours, from injury and started on seizure prophylaxis if they meet the predefined inclusion and exclusion criteria. Patients randomized to the levetiracetam group will receive levetiracetam 1000 mg intravenously or by mouth twice daily for a total of 7 days. Patients randomized to the lacosamide group will receive lacosamide 200 mg intravenously or by mouth twice daily for a total of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosis of moderate to severe traumatic brain injury
* Seizure prophylaxis with one of the two study drugs within 24 hours of initial injury
* Patients admitted into the trauma team service

Exclusion Criteria:

* Enrolled in another interventional drug study
* Any active, witnessed, or unable to rule out seizure prior to prophylaxis initiation
* Received antiseizure medication (ASM), for prophylaxis or treatment, prior to randomization
* History of seizures
* On anti-epileptic medications for seizures or indications other than seizures prior to admission
* Documented history of alcohol withdrawal and experiencing alcohol withdrawal on admission with initiation of clinical institute withdrawal assessment scale revised (CIWA-Ar) or modified Minnesota Detoxification Scale (mMINDS) requiring treatment
* Spinal cord injury (SCI), confirmed by radiographic imaging demonstrating cervical (C1 to C8) or thoracic-spine (T1 to T12) injuries consistent with spinal cord injury
* History of bradycardia or permanent pacemaker or signs of bradycardia with HR < 55 bpm for > 5 min not on medications that cause bradycardia
* End-stage renal disease (ESRD)
* Death, withdrawal of life support or transfer to hospice within 24 hours
* Pregnant or incarcerated
* Baseline GCS < 13 or unable to determine baseline GCS
* Patient with a GCS of 15 or Legally Authorize Representative (LAR) unable to provide informed consent prior to randomization, or unable to read and understand English, Spanish, Vietnamese, Russian, Arabic, or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Early Post-traumatic Seizure | Up to day 7 post injury
  Number of early post-traumatic seizures documented

SECONDARY OUTCOMES:
Richmond Agitation-Sedation Scale Score Attainment | Hour 24, hour 48, day 7 and day 10 post first drug administration
  It will be noted if the participant attains their Richmond Agitation-Sedation Scale (RASS) score goal within the various time periods. Goal scores will vary per participant from -5 to +1, depending on individualized sedation goals. If participants are not maintained within their RASS goal and must receive as-needed or scheduled agitation medications to attain their RASS goal, they will be considered to have agitation.
Administration of Agitation Medications | Hour 24, hour 48, day 7 and day 10
  Use of as needed or scheduled agitation medications
Incidence of Late Post-traumatic Seizures | Day 8 post injury through day 30
  Number of late post-traumatic seizures
Intensive Care Unit Length of Stay | Admission through day 30
  Number of days participant spent in Intensive Care Unit
Number of Readmissions to Intensive Care Unit | Admission through day 30
  Number of times patient is readmitted to the Intensive Care Unit
Total Hospital Length of Stay | Admission through day 30
  Number of days participant was admitted to the hospital
Duration of Mechanical Ventilation | Admission through day 30
  Length of time participant was on mechanical ventilation
Total Cost of Hospitalization | Admission through day 30
  Cost of hospitalization data will be obtained from Surgical Trauma Intensive Care Unit data mart from the Acute Care Surgery Department
Number of In-hospital Mortalities | Admission through day 30
  Number of participant mortalities while admitted to hospital
Post-traumatic Seizure - Operative vs Nonoperative Neurosurgery Management | Admission through day 30
  Of participants who developed a posttraumatic seizure, number of patients who required operative neurosurgery interventions
Post-traumatic Seizure - Subdural Hematoma vs Non-subdural Hematoma | Admission through day 30
  Of participants who developed a posttraumatic seizure, number of patients who had subdural hematomas
Incidence of Agitation Medication Use - Non-intubated Patients | Admission through day 30
  Incidence of agitation medication use (as-needed or scheduled) in non-intubated patients will be assessed via chart review
Post-traumatic Seizure with Anti-Seizure Medication | Day 7
  Number of participants who received anti-seizure medication within four hours vs 5-24 hours from injury

CONTACTS AND LOCATIONS:
Overall Officials: Rita Brintzenhoff, MD, Principal Investigator — Atrium Health Carolina Medical Center
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No